CLINICAL TRIAL: NCT05697835
Title: Behavioral Activation and Medication Optimization for Perioperative Mental Health in Orthopedic Surgery
Brief Title: Perioperative Mental Health in Orthopedic Surgery
Acronym: CPMH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ryan Calfee, MD, Professor of Orthopaedic Surgery, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202301070; P50MH122351 (NIH)
Record Dates: First submitted 2023-01-14; First posted 2023-01-26 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Orthopedic Surgery; Older Adults; Depression; Anxiety
Keywords: Behavioral: Behavioral activation; Medication optimization; Care as usual
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Hybrid Type 1 effectiveness-implementation randomized controlled trial design
Who Masked: Investigator, Outcomes Assessor
Masking Description: Study staff responsible for administering ratings and collecting outcomes throughout the study are blinded. The investigator(s) are also blinded. This blinding is kept throughout the study until data collection is complete. At the end of the follow-up, the study coordinator will complete a blinding question to try to guess the arm to which each participant was allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral activation and medication optimization (Experimental): Behavioral activation (BA) will begin perioperatively and will span across 3 months postoperatively, with sessions approximately weekly or biweekly, depending on patient preference & health condition.
  Medications will be reviewed by a team of interventionists to minimize brain-toxic medications and optimize doses of antidepressants and other mental health medications. In-hospital and after discharge, the interventionists' role will include coordinating with the care teams to ensure that medication changes that were introduced preoperatively are maintained.
  Interventions: Behavioral: Behavioral activation; Other: Medication optimzation
- Control (treatment as usual) (Other): Participants in control arm will continue care as usual. They will receive printed resources for supporting sleep hygiene, stress reduction, cognitive and mental health exercises, as well as community resources for older adults.
  Interventions: Other: Care as usual

INTERVENTIONS:
Behavioral: Behavioral activation — The behavioral intervention will consist of behavioral activation (BA), the basic premise of which is to help people with mental health problems to engage in activities that are reinforcing or meaningful and guided by their personal values
  Arms: Behavioral activation and medication optimization
Other: Medication optimzation — Medication optimization consists of a simple set of principles: reconcile patient's medications, identify the patient's likely need for, and interest in, a medication adjustment, make the adjustment, and assess the response to that adjustment.
  Arms: Behavioral activation and medication optimization
Other: Care as usual — Care as usual, with written resources provided
  Arms: Control (treatment as usual)

SUMMARY:
This Hybrid 1 Study will test the effectiveness of a bundled intervention comprised of behavioral activation and medication optimization in reducing symptoms of depression and anxiety in older adults undergoing Orthopedic surgery (compared with usual care), while examining implementation outcomes.

ELIGIBILITY:
Inclusion criteria:

* Adults ≥ 60 years
* Scheduled primary hip or primary knee arthroplasty procedure
* PHQ-ADS ≥ 10, indicating clinically significant depression or anxiety symptoms

Exclusion criteria:

* Barrier to communication (Unable to read, speak, and understand English)
* Severe cognitive impairment screened by the SBT (Short Blessed Test) >10
* Acutely suicidal
* Previous participation in this study or another CPMH study of the intervention bundle or its feasibility.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2025-03-19 (Actual)

PRIMARY OUTCOMES:
PHQ-ADS | 3 months post-operatively
  PHQ-ADS (Patient Health Questionnaire Anxiety and Depression Scale) scores will be compared between the two study arms 3 months after surgery.
  PHQ-ADS is a composite measure of anxiety and depression. PHQ-ADS scores can range from 0 to 48 (with higher scores indicating more severe depression/anxiety)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Calfee, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holzer KJ, Bartosiak KA, Calfee RP, Hammill CW, Haroutounian S, Kozower BD, Cordner TA, Lenard EM, Freedland KE, Tellor Pennington BR, Wolfe RC, Miller JP, Politi MC, Zhang Y, Yingling MD, Baumann AA, Kannampallil T, Schweiger JA, McKinnon SL, Avidan MS, Lenze EJ, Abraham J. Perioperative mental health intervention for depression and anxiety symptoms in older adults study protocol: design and methods for three linked randomised controlled trials. BMJ Open. 2024 Apr 3;14(4):e082656. doi: 10.1136/bmjopen-2023-082656. PMID 38569683

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-05-29): https://cdn.clinicaltrials.gov/large-docs/35/NCT05697835/SAP_002.pdf